CLINICAL TRIAL: NCT01242436
Title: Whole Body Diffusion MRI for Non-invasive Lesion Detection and Therapy Follow-up: Study With Patients With Ovarian Cancer and Peritoneal Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, katrijn Michielsen, PhD researcher Radiology, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S52920
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Ovarian Cancer; Peritoneal Metastasis
Keywords: Ovarian Cancer; Peritoneal Metastasis; Whole body diffusion MRI; therapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: intravenous contrast administration — The additional burden is restricted to a WB-DWI scan before and during therapy.
  MRI is a technique based on magnetic fields and do not require the use of ionizing radiation. Because of the strong magnetic field, a few precautions should be taken. This means that all metal and magnetized objects must be removed from the patient before entering the MRI room. Patients with a pacemaker, a cardiac defibrillator or other implanted conductor/prosthesis are for this reason not eligible for the study.
  During the examination, an intravenous will be administered. In most cases, patients do not experience any discomfort and the use of this contrast agent is part of the clinical routine.

SUMMARY:
Ovarian cancer is a gynecological cancer with a high risk of mortality. This is because the diagnosis is often been made in an advanced cancer stage with metastases throughout the peritoneum.

An international study led by Prof. Dr. Ignace Vergote (Gynaecological Oncology) showed for the first time that patients in such an advanced stage of ovarian cancer who received first three neoadjuvant platinum-based chemotherapy regimens followed by interval debulking surgery, and in turn followed by at least 3 treatment with platinum-based chemotherapy, had fewer complications than patients treated with primary debulking surgery followed by chemotherapy. Moreover, the final survival rate in both groups seemed to be similar. The most important prognostic marker appeared to be whether patients with primary or interval surgery no longer had a visible residual tumor after the treatment. Patients who had only small metastases in the peritoneum, seemed to be better treated with primary surgery (neoadjuvant Vergote I, et al Chemotherapy or Primary Surgery in Stage IIIC or IV Ovarian Crystallising, N Engl J Med 363 (1910): 943 - 953).

Each patient with suspected advanced ovarian cancer should undergo a preoperative evaluation where they assess which of the two treatments is the best option.

The aim of the study is to assess whole body diffusion weighted imaging (WB-DWI) as a non-invasive method, in patients with confirmed ovarian cancer in the presence of peritoneal metastases. This is to assess which of the two treatments (primary debulking surgery followed chemotherapy versus platinum-based neoadjuvant chemotherapy followed by interval debulking surgery, followed in turn by chemotherapy) is the best option for a particular type of patient.

DETAILED DESCRIPTION:
BACKGROUND OF THE STUDY

Ovarian cancer is a gynecological cancer with a high risk of mortality. This is because the diagnosis is often been made in an advanced cancer stage with metastases throughout the peritoneum. The standard treatment for this condition till now consisted of primary debulking surgery where the tumor, the uterus and both the ovaries were removed, followed by a minimum of six treatments with platinum-based chemotherapy. This operation is often accompanied by serious complications such as for example bleedings, embolic events, infections and in extreme cases, even mortality. An international study led by Prof. Dr. Ignace Vergote (Gynaecological Oncology) showed for the first time that patients in such an advanced stage of ovarian cancer who received first three neoadjuvant platinum-based chemotherapy regimens followed by interval debulking surgery, and in turn followed by at least 3 treatment with platinum-based chemotherapy, had fewer complications than patients treated with primary debulking surgery followed by chemotherapy. Moreover, the final survival rate in both groups seemed to be similar. The most important prognostic marker appeared to be whether patients with primary or interval surgery no longer had a visible residual tumor after the treatment. Patients who had only small metastases in the peritoneum, seemed to be better treated with primary surgery (neoadjuvant Vergote I, et al Chemotherapy or Primary Surgery in Stage IIIC or IV Ovarian Crystallising, N Engl J Med 363 (1910): 943 - 953).

Each patient with suspected advanced ovarian cancer should undergo a preoperative evaluation where they assess which of the two treatments is the best option. This should of course, for each individual patient, take into account comorbidity, cancer stage, number and location of the metastases etc. Currently,[18F] FDG-PET/CT, CT and conventional MRI are being used for staging, detecting recurrence and metastasis and for evaluating therapy response. These techniques have some disadvantages. A PET study takes a long time to perform and makes use of radioactive material. The addition of CT also gives rise to additional radiation. [18F] FDG accumulates in inflammatory cells in the tumor. This can explain the difficulties concerning early evaluation of treatment response. Although CT allows high resolution images of the entire body, sometimes the technology lacks sufficient sensitivity or specificity. Although conventional MRI has the highest sensitivity for detection of liver metastases, the lack of efficient whole-body imaging for staging a disadvantage when assessing systemic tumor spread and metastasis. Small peritoneal metastases are therefore often missed with this technique.

Diffusion-weighted imaging (DWI) is an emerging technology that is currently being uses in cancer imaging. Here the difference in movement of water molecules provides information about the integrity of cellular membranes. DWI has the advantage that no contrast material is required and there is also no need for exposure to ionizing radiation. Further developments in technology allowed for an acceptable time in whole body conducting research, so we should be able to image gastrointestinal tumors with this whole body technique.

AIM OF THE STUDY

The aim of the study is to assess whole body diffusion weighted imaging (WB-DWI) as a non-invasive method, in patients with confirmed ovarian cancer in the presence of peritoneal metastases. This is to assess which of the two treatments (primary debulking surgery followed chemotherapy versus platinum-based neoadjuvant chemotherapy followed by interval debulking surgery, followed in turn by chemotherapy) is the best option for a particular type of patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage IIIC or IV epithelial ovarian cancer in the presence of peritoneal metastasis are, on a voluntary basis, enrolled in the study. These are patients who 'll either underwent primary debulking surgery followed by at least six courses of platinum-based chemotherapy or patients who will be assigned to three courses of neoadjuvant platinum-based chemotherapy followed by interval debulking surgery, followed in turn by at least three courses of platinum-based chemotherapy.

Exclusion Criteria:

* Patients with known contra-indications for MRI (cardiac pacemakers, cochlear implants, claustrophobic patients) will be excluded from this study. And so are patients with contra-indications to Gadolinium-based contrast agents and patients with a known restricted renal function (GFR < 30 ml/min).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of WB-DWI as a noninvasive method to assess which kind of treatment fits best for a particular patient with ovarian cancer in the presence of peritoneal metastasis | 2011-2015 continuously
  The aim of the study is to assess whole body diffusion weighted imaging (WB-DWI)as a non-invasive method, in patients with confirmed ovarian cancer in the presence of peritoneal metastases. This is to evaluate which of the two treatments (primary debulking surgery followed chemotherapy versus platinum-based neoadjuvant chemotherapy followed by interval debulking surgery, followed in turn by chemotherapy) is the best option for a particular type of patient.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Gasthuisberg, Leuven, Leuven, Belgium

REFERENCES:
- See also: Whole-body MRI with diffusion-weighted sequence for staging of patients with suspected ovarian cancer: a clinical feasibility study in comparison to CT and FDG-PET/CT (Eur Radiol) — http://www.ncbi.nlm.nih.gov/pubmed/24322510